CLINICAL TRIAL: NCT03357770
Title: Evaluating the Maximum Tolerated Dose of Mesenchymal Stem Cells From Umbilical
Brief Title: The Maximum Tolerated Dose of Mesenchymal Stem Cells From Umbilical Cord
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, yangziyi, arthritis clinic and research center, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PUPH20170910
Record Dates: First submitted 2017-11-25; First posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Knee Osteoarthritis; Umbilical Cord Bleeding
Keywords: mesenchymal stem cells; Knee Osteoarthritis; Umbilical Cord
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- low dose of mesenchymal stem cells (Experimental): Three groups of patients were enrolled in this study. Every group includes three patients. The three groups of patients were treated with high, medium and low dose of cytokine.The low-dose is 1 × 10^7cells / 3mL
  Interventions: Drug: mesenchymal stem cells
- medium dose of mesenchymal stem cells (Experimental): the medium-dose is 5 × 10^7cells / 3mL
  Interventions: Drug: mesenchymal stem cells
- high dose of mesenchymal stem cells (Experimental): the high dose is 1 × 10^8cells / 3mL
  Interventions: Drug: mesenchymal stem cells

INTERVENTIONS:
Drug: mesenchymal stem cells — we will enroll three groups of patients, and they will be therapized by high, medium, and low-dose cytotoxic respectively to evaluate the dose-limiting toxicity (DLT) and establish the maximum tolerated dose (MTD). Dose and cell concentration selection will be based on previous literature [5]. The low-dose is 1 × 10^7cells / 3mL, the medium-dose is 5 × 10^7cells / 3mL and the high dose is 1 × 10^8cells / 3mL

SUMMARY:
The aim of this study was to evaluate the maximum tolerated dose of Mesenchymal Stem Cells (MSCs) from umbilical cord in the treatment of human knee OA

DETAILED DESCRIPTION:
This is a single-centre, quadruple blined, randomized controlled trail with a total of 9 knee osteoarthrits patients as participants, who will be randomly assigned into high dose group, moderate dose group or low dose group. The participants in the high dose group will receive the treatment of high dose MSCs (1×10^8cells/3mL) anticular injection.The dose of the MSCs in medium dose group is 5×10^7cells/3mL, and the dose in the low dose group is 1×10^7cells/3mL. Unexplained local and systemic symptoms will be assessed to determine the the maximum tolerated dose of mesenchymal stem cells in anticular injection.

ELIGIBILITY:
Inclusion Criteria:

① K / L score of 2-3; ② chronic knee pain; ③ no local or systemic infection; ④ without obvious contraindication of the joint puncture from hematology and biochemical tests; ⑤ informed consent. -

Exclusion Criteria:

① older than 75 years old or less than 18 years old, or without full capacity for civil conduct; ② HIV, hepatitis virus or syphilis virus infection or their serology is positive; ③ BMI index is greater than 30; ④ congenital or acquired knee deformity; ⑤ pregnant or lactating women; ⑥ tumor patients; ⑦ immunodeficiency patients; ⑧ intra-articular drug injection history within 3 months; ⑨ participating in other clinical trials; ⑩ other patients who researchers believe are not eligible for inclusion such as suffering from other concomitant diseases.-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Unexplained local and systemic symptoms or death | 6 months
  The severity of AE must be recorded and graded according to the CTCAE criteria, and its relationship to therapy must be assessed according to the following definition:①not related: there is evidence that the cause of adverse events is not due to intra-articular injection therapy (such as previous conditions, potential diseases, concurrent diseases); ②related: AE and intra-articular injection are time-related and it is known or suspected that intra-articular injection of drugs can cause the AE; ③it can't be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Jianhao Lin, MD, Principal Investigator — arthritis clinic and research center

IPD SHARING:
Plan to Share IPD: No